CLINICAL TRIAL: NCT01161212
Title: Physical Activity, Health-related Quality of Life and Corpulence Among French Schoolchildren
Brief Title: REGULarity of Physical ActivitieS (REGUL'APS)
Acronym: REGUL'APS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nancy (Other)
Collaborators: IVRSP: Institut Virtuel de Recherche en Santé Publique (Unknown)
Responsible Party: Anne Vuillemin, PhD, Public Health School, Laboratory EA4360 Apemac
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Regulaps2006; CNIL n°05-1340 (Other: French Data Protection Authority); CCTIRS-05.65 (Other: National Consultative Ethics Committee for Health and Life Sciences)
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-07

CONDITIONS: Overweight; Obesity
Keywords: body mass index; health-related quality of life; physical education; children; cluster randomized controlled trial; prevention; Child; French; Schoolchildren
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Other)
  Interventions: Other: Physical education sessions
- Intervention group (Other)
  Interventions: Other: Physical education sessions

INTERVENTIONS:
Other: Physical education sessions — 3(60 minutes each) or 4 (45 minutes each) short sessions of physical education (PE) sessions
  Arms: Intervention group
Other: Physical education sessions — 1 (3 hours) or 2 long PE sessions (1 hour and 30 minutes each)
  Arms: Control group

SUMMARY:
In French primary schools, children participate in 3 compulsory hours of physical education (PE) each week unless they have a medical contra-indication. But, there is no scientific evidence (randomized trial) that a weekly physical activity splitting up of these 3 hours of PE brings or not the same effects, particularly to prevent overweight or obesity.

Regul'aps is a cluster randomized controlled trial which wants to evaluate whether splitting up the 3 hours into 3 or 4 sessions (vs. 1-2 sessions) of PE per week has an effect on speed of a BMI increase and on health-related quality of life (HRQoL) over the school year.

Study hypothesis: reduction of speed of increase of BMI and an increase of HRQoL

ELIGIBILITY:
Inclusion Criteria:

* All teachers under the cover of the headmasters in charge of classes from grades 2 to 5 in 2 counties in the Lorraine region of France (Meurthe-et-Moselle and Vosges [District of Golbey])
* headmasters or teachers had to agree to modify the organisation of PE sessions

Exclusion Criteria:

* Classes composed only of 2d grade
* Set schedule of physical educational sessions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2005-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) and waist circumference | September 2006 and June 2007
  September 2006 : at the beginning of school year June 2007 : at the end of school year (31 weeks later)

SECONDARY OUTCOMES:
Health-related quality of life | September 2006 and June 2007
  September 2006 : at the beginning of school year June 2007 : at the end of school year (31 weeks later)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Vuillemin, PhD, Principal Investigator — Public Health School, Laboratory EA4360 Apemac
Locations (1):
- Public health School, Laboratory EA4360 Apemac, Vandœuvre-lès-Nancy, France